CLINICAL TRIAL: NCT06095674
Title: ImmunoTHerapy Adjacent to Cervical CAncer (ITHACA) Study: Safety, Toxicity and Immunological Effects of Peritumorally Delivered Immunotherapy in Early-stage Cervical Cancer
Brief Title: ImmunoTHerapy Adjacent to Cervical CAncer (ITHACA) Study
Acronym: ITHACA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Cancer Society (Other); Agenus Inc. (Industry)
Responsible Party: Principal Investigator, C.H. (Stijn) Mom, Principle investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14244
Record Dates: First submitted 2023-09-04; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Cervical Cancer
Keywords: Immune therapy; Check point inhibitor; Peritumoral administration
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 checkpoint inhibitor and CTLA-4 inhibitor (Experimental): Both antibodies will be peritumorally administered in early-stage cervical cancer prior to surgery.
  Interventions: Drug: Anti-PD-1 antibody balstilimab

INTERVENTIONS:
Drug: Anti-PD-1 antibody balstilimab — Both antibodies will be neoadjuvantly administered around the cervical tumor.
  Other Names: Anti-CTLA-4 antibody botensilimab

SUMMARY:
The ITHACA study is a phase I study evaluating the safety and toxicity of a peritumorally injected PD-1 checkpoint inhibitor, in combination with a multifunctional CTLA-4 inhibitor, in early-stage cervical cancer.

DETAILED DESCRIPTION:
In this single arm, open label phase I study, the investigators will study the safety and toxicity of the combination of a PD-1 checkpoint inhibitor and a multifunctional CTLA-4 inhibitor when injected peritumorally prior to surgery in early-stage cervical cancer. Additional objectives are to describe dose limiting toxicities, to determine the maximum tolerated doses and to study the effects on the tumor and lymph node microenvironment, and on immune subsets in peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* early-stage cervical cancer
* scheduled for (radical) hysterectomy and pelvic lymph node dissection

Exclusion Criteria:

* previous treatment with checkpoint inhibitors
* use of immunosuppressive medication within 28 days of the injection of the study medication
* history of other malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | 2 years
  Type and severity of side effects according to CTCAE v 5.0.

SECONDARY OUTCOMES:
Maximum tolerated dose | 2 years
  The highest dose administered without unacceptable toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Constantijne H Mom, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands